CLINICAL TRIAL: NCT06249945
Title: The Safety and Efficacy of Empagliflozin in Patients With End-stage Renal Disease and Heart Failure With Preserved Ejection Fraction - a Randomized Controlled Trial
Brief Title: EMPAgliflozin in Heart Failure With PReserved Ejection Fraction and End Stage Renal Disease
Acronym: EMPA-PRED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301126MINC
Record Dates: First submitted 2024-01-21; First posted 2024-02-08 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction; End Stage Renal Disease on Dialysis
Keywords: end-stage renal disease; sodium-glucose co-transporter 2 inhibitors; heart failure; diastolic function; empagliflozin
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- empagliflozin (Experimental): Jardiance, 25 mg, QD, for 6 months
  Interventions: Drug: Empagliflozin 25 MG
- Placebo (Placebo Comparator): QD, for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — The medication will be packed in a customized sealed jar and labeled on the exterior of the jar.
  Other Names: Jardiance 25 MG
  Arms: empagliflozin
Drug: Placebo — The placebo tablet is manufactured by Prince Pharmaceutical Co., Ltd, a leading manufacturer of nutritional supplements with certifications including cGMP, GMP, ISO, and HACCP. The Prince Pharmaceutical also provides Original Equipment Manufacturing (OEM)/Original Design Manufacturing (ODM) services for a wide array of tablet shapes, and post-processing techniques such as film coating and sugar coating.
  Arms: Placebo

SUMMARY:
The presence of CKD has been linked to the development of HFpEF. Currently, the treatment for HFpEF is limited. SGLT2i are one of the few drug classes that have proven efficacy in HFpEF in randomized controlled trials. The results of mechanistic studies suggest that the benefits of SGLT2i on diastolic heart failure are independent of their glycosuric actions and may still be present in anuric subjects. Despite the significance of HFpEF in patients with CKD, patients with advanced kidney disease have been excluded from studies investigating anti-heart failure drugs. The effects of SGLT2i in patients under maintenance dialysis are largely unknown. Past pharmacokinetics and pharmacodynamics studies on empagliflozin in patients with end-stage renal disease (ESRD) demonstrated that the use of empagliflozin in patients with ESRD seemed safe, yet its efficacy remains to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old
* ESRD under chronic, maintenance dialysis with stable dry weight for the past 6 months
* Prior diagnosis of HFpEF, as defined by a score of ≥5 on the HFA-PEFF diagnostic algorithm.

Exclusion Criteria:

* Age <20 years old
* Ongoing pregnancy
* NYHA class IV heart failure
* Any hospitalization for heart failure within the past month Ongoing acute urinary tract infection at the time of screening
* Known acute genital infection
* Severe peripheral artery disease (Rutherford category 4-6)
* Acute coronary syndrome, stroke or transient ischemic attack within the past month
* Recent initiation of chronic maintenance hemodialysis within 6 months
* Adjustment of dry weight with changes greater than 5% of body weight within the past month
* Documented left ventricular ejection fraction =<40% by any imaging modality within 1 month of screening
* Refused informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitral early (E) and late (A) diastolic filling velocity ratio (E/A) | 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day

SECONDARY OUTCOMES:
LV end-systolic volume index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LV end-diastolic volume index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LA volume index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LV ejection fraction | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Left ventricular mass index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Global longitudinal strain | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LA strain | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Mitral inflow deceleration time | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Mitral inflow deceleration time LV relative wall thickness | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Tricuspid regurgitation peak gradient (TRPG) | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
NT-proBNP | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
HbA1c | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
Lipid profile | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
KCCQ-OS | 12 weeks and 24 weeks of treatment
  Performed on non-dialysis day
6-minute walking distance | 12 weeks and 24 weeks of treatment
  Performed on non-dialysis day
3-minute heart rate variability | 12 weeks and 24 weeks of treatment
  During hemodialysis session
Blood pressure | 12 weeks and 24 weeks of treatment
  Obtained pre-dialysis session
Major adverse cardiovascular events (composite of CV death, myocardial infarction, stroke) | 24 weeks of treatment
  By medical record confirmation and by interview
Lower extremity non-traumatic amputation or revascularization | 24 weeks of treatment
  By medical record confirmation and by interview
All-cause mortality | 24 weeks of treatment
  By medical record confirmation and by interview
Hospitalization for heart failure | 24 weeks of treatment
  By medical record confirmation and by interview
Hypoglycemic events | 24 weeks of treatment
  By medical record confirmation and by interview
Diabetic ketoacidosis | 24 weeks of treatment
  By medical record confirmation and by interview
Urinary tract infection | 24 weeks of treatment
  By medical record confirmation and by interview
Genital tract infection | 24 weeks of treatment
  By medical record confirmation and by interview
Hypokalemia | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session

CONTACTS AND LOCATIONS:
Overall Officials: Donna SH Lin, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital; Chih-Cheng Wu, MD. PhD, Principal Investigator — National Taiwan University Hsin-Chu Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital Hsinchu Branch, Hsinchu
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] Kalantar-Zadeh K, Jafar TH, Nitsch D, Neuen BL, Perkovic V. Chronic kidney disease. Lancet. 2021 Aug 28;398(10302):786-802. doi: 10.1016/S0140-6736(21)00519-5. Epub 2021 Jun 24. PMID 34175022
- [Background] Ronco C, Haapio M, House AA, Anavekar N, Bellomo R. Cardiorenal syndrome. J Am Coll Cardiol. 2008 Nov 4;52(19):1527-39. doi: 10.1016/j.jacc.2008.07.051. PMID 19007588
- [Background] Bansal N, Zelnick L, Bhat Z, Dobre M, He J, Lash J, Jaar B, Mehta R, Raj D, Rincon-Choles H, Saunders M, Schrauben S, Weir M, Wright J, Go AS; CRIC Study Investigators. Burden and Outcomes of Heart Failure Hospitalizations in Adults With Chronic Kidney Disease. J Am Coll Cardiol. 2019 Jun 4;73(21):2691-2700. doi: 10.1016/j.jacc.2019.02.071. PMID 31146814
- [Background] Kotecha D, Gill SK, Flather MD, Holmes J, Packer M, Rosano G, Bohm M, McMurray JJV, Wikstrand J, Anker SD, van Veldhuisen DJ, Manzano L, von Lueder TG, Rigby AS, Andersson B, Kjekshus J, Wedel H, Ruschitzka F, Cleland JGF, Damman K, Redon J, Coats AJS; Beta-Blockers in Heart Failure Collaborative Group. Impact of Renal Impairment on Beta-Blocker Efficacy in Patients With Heart Failure. J Am Coll Cardiol. 2019 Dec 10;74(23):2893-2904. doi: 10.1016/j.jacc.2019.09.059. PMID 31806133
- [Background] Ferro CJ, Mark PB, Kanbay M, Sarafidis P, Heine GH, Rossignol P, Massy ZA, Mallamaci F, Valdivielso JM, Malyszko J, Verhaar MC, Ekart R, Vanholder R, London G, Ortiz A, Zoccali C. Lipid management in patients with chronic kidney disease. Nat Rev Nephrol. 2018 Dec;14(12):727-749. doi: 10.1038/s41581-018-0072-9. PMID 30361677
- [Background] Shah KS, Fang JC. Is Heart Failure with Preserved Ejection Fraction a Kidney Disorder? Curr Hypertens Rep. 2019 Oct 10;21(11):86. doi: 10.1007/s11906-019-0993-0. PMID 31599363
- [Background] Ter Maaten JM, Damman K, Verhaar MC, Paulus WJ, Duncker DJ, Cheng C, van Heerebeek L, Hillege HL, Lam CS, Navis G, Voors AA. Connecting heart failure with preserved ejection fraction and renal dysfunction: the role of endothelial dysfunction and inflammation. Eur J Heart Fail. 2016 Jun;18(6):588-98. doi: 10.1002/ejhf.497. Epub 2016 Feb 10. PMID 26861140
- [Background] Cohen JB, Schrauben SJ, Zhao L, Basso MD, Cvijic ME, Li Z, Yarde M, Wang Z, Bhattacharya PT, Chirinos DA, Prenner S, Zamani P, Seiffert DA, Car BD, Gordon DA, Margulies K, Cappola T, Chirinos JA. Clinical Phenogroups in Heart Failure With Preserved Ejection Fraction: Detailed Phenotypes, Prognosis, and Response to Spironolactone. JACC Heart Fail. 2020 Mar;8(3):172-184. doi: 10.1016/j.jchf.2019.09.009. Epub 2020 Jan 8. PMID 31926856
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- [Background] Verma S, Mazer CD, Yan AT, Mason T, Garg V, Teoh H, Zuo F, Quan A, Farkouh ME, Fitchett DH, Goodman SG, Goldenberg RM, Al-Omran M, Gilbert RE, Bhatt DL, Leiter LA, Juni P, Zinman B, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease: The EMPA-HEART CardioLink-6 Randomized Clinical Trial. Circulation. 2019 Nov 19;140(21):1693-1702. doi: 10.1161/CIRCULATIONAHA.119.042375. Epub 2019 Aug 22. PMID 31434508
- [Background] Ersboll M, Jurgens M, Hasbak P, Kjaer A, Wolsk E, Zerahn B, Brandt-Jacobsen NH, Gaede P, Rossing P, Faber J, Inzucchi SE, Gustafsson F, Schou M, Kistorp C. Effect of empagliflozin on myocardial structure and function in patients with type 2 diabetes at high cardiovascular risk: the SIMPLE randomized clinical trial. Int J Cardiovasc Imaging. 2022 Mar;38(3):579-587. doi: 10.1007/s10554-021-02443-5. Epub 2021 Oct 20. PMID 34669059
- [Background] Soga F, Tanaka H, Tatsumi K, Mochizuki Y, Sano H, Toki H, Matsumoto K, Shite J, Takaoka H, Doi T, Hirata KI. Impact of Dapagliflozin on the Left Ventricular Diastolic Function in Diabetic Patients with Heart Failure Complicating Cardiovascular Risk Factors. Intern Med. 2021;60(15):2367-2374. doi: 10.2169/internalmedicine.6127-20. Epub 2021 Aug 1. PMID 34334588
- [Background] Li X, Lu Q, Qiu Y, do Carmo JM, Wang Z, da Silva AA, Mouton A, Omoto ACM, Hall ME, Li J, Hall JE. Direct Cardiac Actions of the Sodium Glucose Co-Transporter 2 Inhibitor Empagliflozin Improve Myocardial Oxidative Phosphorylation and Attenuate Pressure-Overload Heart Failure. J Am Heart Assoc. 2021 Mar 16;10(6):e018298. doi: 10.1161/JAHA.120.018298. Epub 2021 Mar 13. PMID 33719499
- [Background] Pabel S, Wagner S, Bollenberg H, Bengel P, Kovacs A, Schach C, Tirilomis P, Mustroph J, Renner A, Gummert J, Fischer T, Van Linthout S, Tschope C, Streckfuss-Bomeke K, Hasenfuss G, Maier LS, Hamdani N, Sossalla S. Empagliflozin directly improves diastolic function in human heart failure. Eur J Heart Fail. 2018 Dec;20(12):1690-1700. doi: 10.1002/ejhf.1328. Epub 2018 Oct 17. PMID 30328645
- [Background] Macha S, Mattheus M, Halabi A, Pinnetti S, Woerle HJ, Broedl UC. Pharmacokinetics, pharmacodynamics and safety of empagliflozin, a sodium glucose cotransporter 2 (SGLT2) inhibitor, in subjects with renal impairment. Diabetes Obes Metab. 2014 Mar;16(3):215-22. doi: 10.1111/dom.12182. Epub 2013 Aug 19. PMID 23859488
- [Background] Pieske B, Tschope C, de Boer RA, Fraser AG, Anker SD, Donal E, Edelmann F, Fu M, Guazzi M, Lam CSP, Lancellotti P, Melenovsky V, Morris DA, Nagel E, Pieske-Kraigher E, Ponikowski P, Solomon SD, Vasan RS, Rutten FH, Voors AA, Ruschitzka F, Paulus WJ, Seferovic P, Filippatos G. How to diagnose heart failure with preserved ejection fraction: the HFA-PEFF diagnostic algorithm: a consensus recommendation from the Heart Failure Association (HFA) of the European Society of Cardiology (ESC). Eur Heart J. 2019 Oct 21;40(40):3297-3317. doi: 10.1093/eurheartj/ehz641. PMID 31504452
- [Background] Rau M, Thiele K, Hartmann NK, Schuh A, Altiok E, Mollmann J, Keszei AP, Bohm M, Marx N, Lehrke M. Empagliflozin does not change cardiac index nor systemic vascular resistance but rapidly improves left ventricular filling pressure in patients with type 2 diabetes: a randomized controlled study. Cardiovasc Diabetol. 2021 Jan 7;20(1):6. doi: 10.1186/s12933-020-01175-5. PMID 33413355
- [Background] Shim CY, Seo J, Cho I, Lee CJ, Cho IJ, Lhagvasuren P, Kang SM, Ha JW, Han G, Jang Y, Hong GR. Randomized, Controlled Trial to Evaluate the Effect of Dapagliflozin on Left Ventricular Diastolic Function in Patients With Type 2 Diabetes Mellitus: The IDDIA Trial. Circulation. 2021 Feb 2;143(5):510-512. doi: 10.1161/CIRCULATIONAHA.120.051992. Epub 2020 Nov 13. No abstract available. PMID 33186508
- [Background] Junger C, Prochaska JH, Gori T, Schulz A, Binder H, Daiber A, Koeck T, Rapp S, Lackner KJ, Munzel T, Wild PS. Rationale and design of the effects of EMpagliflozin on left ventricular DIAstolic function in diabetes (EmDia) study. J Cardiovasc Med (Hagerstown). 2022 Mar 1;23(3):191-197. doi: 10.2459/JCM.0000000000001267. PMID 34939776
- [Background] Jurgens M, Schou M, Hasbak P, Kjaer A, Wolsk E, Zerahn B, Wiberg M, Brandt NH, Gaede PH, Rossing P, Faber J, Inzucchi S, Gustafsson F, Kistorp CM. Design of a randomised controlled trial of the effects of empagliflozin on myocardial perfusion, function and metabolism in type 2 diabetes patients at high cardiovascular risk (the SIMPLE trial). BMJ Open. 2019 Nov 27;9(11):e029098. doi: 10.1136/bmjopen-2019-029098. PMID 31780586
- [Derived] Lin DS, Lo HY, Yang CW, Wu CC. Safety and Short-Term Effects of Empagliflozin in Patients with Heart Failure and End-Stage Renal Disease. Am J Cardiovasc Drugs. 2025 Aug 25. doi: 10.1007/s40256-025-00760-x. Online ahead of print. PMID 40855136